CLINICAL TRIAL: NCT05870748
Title: REFRaME-O1: A Phase 2/3 Open-label Study Evaluating the Efficacy and Safety of Luveltamab Tazevibulin (STRO-002) Versus Investigator's Choice (IC) Chemotherapy in Women With Relapsed Platinum-resistant Epithelial Ovarian Cancer (Including Fallopian Tube or Primary Peritoneal Cancers) Expressing Folate Receptor Alpha (FOLR1)
Brief Title: REFRaME-O1: A Study to Investigate the Efficacy and Safety of Luveltamab Tazevibulin Versus Investigator's Choice (IC) Chemotherapy in Women With Ovarian Cancer (Including Fallopian Tube or Primary Peritoneal Cancers) Expressing FOLR1
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to strategic business considerations, Sutro has deprioritized the development of luveltamab tazevibulin, leading to termination of the REFRaME program. This decision is not related to any safety or efficacy concerns associated with luvelta
Sponsor: Sutro Biopharma, Inc. (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Asia-Pacific Gynecologic Oncology Trials Group (APGOT) (Unknown); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRO-002-GM3; GOG-3086 (Other: GOG Foundation); ENGOT-OV79 (Other: European Network of Gynaecological Oncological Trial Groups); GEICO-134-O (Other: European Network of Gynaecological Oncological Trial Groups); APGOT-OV9 (Other: Asia-Pacific Gynecologic Oncology Trials Group)
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Platinum-resistant Ovarian Cancer
Keywords: FOLR1; FolRα; FRα; folate receptor alpha; antibody drug conjugate; Luveltamab tazevibulin; STRO-002; luvelta
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — pegfilgrastim; Gemcitabine; Paclitaxel; liposomal doxorubicin; Topotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Luveltamab tazevibulin dose Cohort A (Experimental): 5.2 mg/kg q3w with prophylactic pegfilgrastim for 2 cycles followed by 4.3 mg/kg q3w for Cycle 3 onwards
  Interventions: Drug: Luveltamab tazevibulin; Drug: Pegfilgrastim
- Luveltamab tazevibulin dose Cohort B (Experimental): 4.3 mg/kg q3w
  Interventions: Drug: Luveltamab tazevibulin
- Part 2: IC Chemotherapy (Active Comparator): * Gemcitabine 1000 mg/m2 on Days 1, 8, and 15 q4w or 1000mg/m2 on Days 1 and 8 q3w
  * Paclitaxel 80 mg/m2 on Days 1, 8, and 15 q4w
  * Pegylated Liposomal Doxorubicin (PLD) 40 mg/m2 q4w
  * Topotecan 4.0 mg/m2on Day 1, 8, and 15 q4w or 1.25 mg/m2 on Days 1 - 5 q3w
  Interventions: Drug: Gemcitabine; Drug: Paclitaxel; Drug: Pegylated liposomal doxorubicin; Drug: Topotecan

INTERVENTIONS:
Drug: Luveltamab tazevibulin — Luveltamab tazevibulin is an antibody-drug conjugate targeting FOLR1. It consists of an IgG1 antibody (SP8166) conjugated to cleavable 3-3-aminophenyl hemiasterlin drug-linkers at 4 sites. The active warhead (SC209) inhibits tubulin polymerization leading to mitotic arrest and cell death.
  Other Names: STRO-002; Luvelta
  Arms: Luveltamab tazevibulin dose Cohort A; Luveltamab tazevibulin dose Cohort B
Drug: Pegfilgrastim — Pegfilgrastim or pegylated G-CSF is approved and used to decrease the incidence of infection in patients receiving myelosuppressive anti-cancer drugs. It increases the proliferation and differentiation of neutrophils.
  Other Names: Neulasta
  Arms: Luveltamab tazevibulin dose Cohort A
Drug: Gemcitabine — Gemcitabine is a chemotherapy regimen used for treating platinum-resistant ovarian cancer. It inhibits ribonucleotide reductase and DNA polymerase, hindering tumor cell growth and promoting cell death.
  Arms: Part 2: IC Chemotherapy
Drug: Paclitaxel — Paclitaxel is a chemotherapy regimen approved for treatment of previously treated ovarian cancer. It stabilizes microtubules, inhibiting tumor cell replication.
  Arms: Part 2: IC Chemotherapy
Drug: Pegylated liposomal doxorubicin — Pegylated liposomal doxorubicin is a chemotherapy regimen approved for treating platinum-resistant ovarian cancer. It inhibits DNA and RNA synthesis by intercalating between base pairs, obstructing tumor cell division.
  Arms: Part 2: IC Chemotherapy
Drug: Topotecan — Topotecan is a chemotherapy regimen approved for treatment of metastatic ovarian cancer after disease progression on or after initial or subsequent chemotherapy. It binds to topoisomerase I inducing DNA breaks and subsequent tumor cell apoptosis.
  Arms: Part 2: IC Chemotherapy

SUMMARY:
A Phase 2/3 study to investigate the efficacy and safety of luveltamab tazevibulin versus IC chemotherapy in women with ovarian cancer (including fallopian tube or primary peritoneal cancers) expressing FOLR1.

DETAILED DESCRIPTION:
This is a randomized, multicenter, international, open-label, 2-part, Phase 2/3 study designed to assess the efficacy and safety of luveltamab tazevibulin versus IC chemotherapy in subjects with relapsed platinum-resistant epithelial ovarian cancer expressing FOLR1.

Part 1 will consist of 2 luveltamab tazevibulin dosing cohorts (Cohort A and Cohort B), with subjects randomized 1:1. Part 1 will be used to select the optimized dosing regimen.

Part 2 will further evaluate the efficacy and safety of the selected dosing regimen versus IC chemotherapy.

Luveltamab tazevibulin will be administered intravenously (IV) over a 1-hour infusion time every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. High grade serous epithelial ovarian cancer, fallopian tube or primary peritoneal cancer
2. Age ≥ 18 years
3. ECOG performance status 0 to 1
4. Positive FOLR1 expression per central laboratory testing
5. Relapsed platinum-resistant epithelial ovarian cancer and received a total of 1 to 3 prior regimens
6. Prior bevacizumab treatment is required, if labeled and available as standard of care per institutional guidelines, unless subject has documented contraindication
7. At least 1 measurable target lesion per RECIST v1.1
8. Adequate organ function

Exclusion Criteria:

1. Low grade (Grade 1) ovarian carcinoma, clear cell, mucinous, endometrioid, sarcomatous, and mixed histology ovarian carcinomas
2. Prior treatment with a FOLR1- targeting ADCs or with ADCs that contain a tubulin inhibitor
3. Primary platinum-refractory disease
4. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy or to antibody-related fusion protein treatment
5. Pre-existing clinically significant ocular disorders, severe chronic obstructive pulmonary disease or asthma, clinically significant cardiac or cerebrovascular disease, or other significant concurrent, uncontrolled medical condition
6. Previous solid organ transplantation
7. History or clinical signs of meningeal or active central nervous system involvement
8. Concurrent participation in another therapeutic treatment trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months
  time between the date of first dose and the first date of documented progression or death
Objective Response Rate (ORR) | up to 24 months
  Best response of complete response (CR) or partial response (PR) per RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 24 months
  Time between date of first dose and date of death due to an cause or end of study.
Duration of Response (DOR) | up to 24 months
  Confirmed CR or PR from the first documented response to the date of documented disease progression or death.
Incidence and severity of adverse events [Safety and tolerability] | up to 24 months
  Incidence and severity of adverse events (AEs) and clinical laboratory abnormalities.
Quality of life (QLQ-OV28) | up to 24 months
  Quality of Life Questionnaire Ovarian Cancer 28 is a 28-item ovarian cancer supplemental module that evaluates the quality of life of ovarian cancer patients. It assesses abdominal/gastrointestinal symptoms, peripheral neuropathy, other chemotherapy side-effects, hormonal/menopausal symptoms, body image, attitude to disease/treatment and sexual functioning.

CONTACTS AND LOCATIONS:
Locations (63):
- United States (37):
  - Arizona Oncology Associates, PC-Hope, Tucson, Arizona
  - Sutter Health, Daly City, California
  - Scripps Health, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Health South Florida (BHSF) - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - USF Research & Innovation, Tampa, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Nancy N. and J.C. Lewis Cancer & Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Optimum Clinical Research Group, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - Pitt County Memorial Hospital, Inc. ECU Medical Center, Greenville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University Center, Columbus, Ohio
  - Kettering Health, Kettering, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Oklahoma Cancer Specialists and Research Institute- Tulsa Cancer Center, Tulsa, Oklahoma
  - Oncology Associates of Oregon, PC, Eugene, Oregon
  - Providence Gynecologic Oncology Clinic, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sidney Kimmel Cancer Center, Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Texas Oncology-DFW, Dallas, Texas
  - Texas Oncology-San Antonio, San Antonio, Texas
  - Baylor Scott & White Medical Center - Temple (Temple Clinic), Temple, Texas
  - Texas Oncology - The Woodlands, The Woodlands, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Mason Medical Center - Digestive Disease Institute - Liver Center, Seattle, Washington
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Canada (3):
  - McGill University Health Centere (MUHC)-Glen Site, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec (CHUQ) - L'Hotel Dieu de Quebec, Québec, Quebec
  - Princess Margaret Cancer Center, Toronto
- Israel (7):
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - The Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Health New Zealand - Te Whatu Ora Capital, Coast, and Hutt Valley - Wellington Regional Hospital, Newtown, Wellington Region, New Zealand
- Singapore (3):
  - Curie Centre, Oncology centre, Novena
  - National University Cancer Institute (NCIS), Pasir Panjang
  - National Cancer Center Singapore, Singapore
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Gyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Yonsei University, Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No